CLINICAL TRIAL: NCT00265395
Title: A Study to Assess Treatment With PEG-Intron® and Rebetol® in Naïve Patients With Genotype 1 Chronic Hepatitis C and Slow Virological Response
Brief Title: Extended Treatment With PEG-Intron® and Rebetol® in Patients With Genotype 1 Chronic Hepatitis C and Slow Virologic Response (Study P03685)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03685; SUCCESS
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy (Active Comparator): Slow responders (defined as being polymerase chain reaction [PCR] positive at Week 12 with at least 2 log reduction in viral load and PCR negative at Week 24) who are randomized at Week 48 to stop treatment at Week 48.
  Interventions: Drug: Combination of pegylated interferon alfa-2b (PEG-Intron®) and ribavirin (Rebetol®)
- Extended therapy (Experimental): Slow responders (defined as being PCR positive at Week 12 with at least 2 log reduction in viral load and PCR negative at Week 24) who are randomized at Week 48 to continue treatment to Week 72.
  Interventions: Drug: Combination of pegylated interferon alfa-2b and ribavirin

INTERVENTIONS:
Drug: Combination of pegylated interferon alfa-2b (PEG-Intron®) and ribavirin (Rebetol®) — 1. Powder for injection in vial or Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for 48 weeks
  2. 200 mg capsules, oral, weight based dose of 800-1400 mg, daily for 48 weeks
  Other Names: (a) SCH 54031; PEG-Intron; PegIntron; ViraferonPeg.; (b) SCH 18908; Rebetol; REBETOL.
  Arms: Standard therapy
Drug: Combination of pegylated interferon alfa-2b and ribavirin — 1. Powder for injection in vial or Redipen (50, 80, 100, 120, and 150 microgram strength), subcutaneous, dose of 1.5 micrograms/kg, weekly for 72 weeks.
  2. 200 mg capsules, oral, weight based dose of 800-1400 mg, daily for 72 weeks
  Other Names: (a) SCH 54031; PEG-Intron; PegIntron; ViraferonPeg.; (b) SCH 18908; Rebetol; REBETOL.
  Arms: Extended therapy

SUMMARY:
This is a controlled, randomized, parallel-groups, open-label, multinational study designed to evaluate the efficacy and safety of PEG-Intron® (pegylated interferon alfa-2b) plus Rebetol® (ribavirin) in subjects with chronic hepatitis C. It is designed to evaluate whether 72 weeks of treatment with PEG-Intron plus Rebetol is more effective than 48 weeks of treatment in subjects with Genotype 1 chronic hepatitis C who exhibit a slow response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 to 70 years, of either sex.
* Genotype-1 hepatitis C virus (HCV)-ribonucleic acid (RNA)-positive subjects.
* Subjects must be willing to give written informed consent and able to adhere to dosing and visit schedules.
* Confirmation of liver biopsy availability: Availability of a liver biopsy performed within 18 months prior to the Screen visit, with a pathology report confirming the histological diagnosis of chronic hepatitis or liver cirrhosis.
* Compensated liver disease with the following minimum hematological, biochemical, and serological criteria at the screen visit (WNL = within normal limits, ULN = Upper Limit Normal):

  * Hemoglobin values of equal or more than 12 g/dL for females and 13 g/dL for males.
  * White blood cells (WBCs) equal to or more than 3,000/mm^3
  * Neutrophil count equal to or more than 1,500/mm^3
  * Platelet count equal to or more than 80,000/mm^3
  * Direct bilirubin up to 10% above ULN is acceptable.
  * Indirect bilirubin up to 10% above ULN is acceptable (unless non-hepatitis related factors such as Gilbert's disease explain an indirect bilirubin rise). In such cases indirect bilirubin should be less than or equal to 3.0 mg/dL (less than or equal to 51.3 µmol/L)
  * Albumin up to 10% above ULN is acceptable.
  * Serum creatinine up to 10% above ULN is acceptable.
  * Alanine aminotransferase (ALT) level above ULN at Screen.
* At the Screen Visit, fasting glucose must be 70-140 mg/dL. Results between 116-140 mg/dL require repeat fasting glucose to be less than 140 mg/dL and HbA1C less than or equal to 8.5%. HbA1C must be less than or equal to 8.5% in diabetic subjects (whether on medication or diet controlled).
* Antinuclear antibodies (ANA) must be less than or equal to 1:320.
* Thyroid Stimulating Hormone (TSH) WNL whether in euthyroid subjects or subjects requiring medical treatment. (subjects requiring medication to maintain TSH levels within normal limits are eligible if all other inclusion/exclusion criteria are met).
* Confirmation by the principal investigator or a sub-investigator that sexually active females of childbearing potential are practicing adequate contraception.
* Female subjects cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile or using 2 methods of birth control. While abstinence from sexual activity is the only certain method to prevent pregnancy, female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use a combination of the following 2 methods :

  * Contraceptive pill or intrauterine device (IUD) or depot hormonal preparation (ring, injection implant) and
  * A barrier method of contraception such as diaphragm, sponge with spermicide, condom, or a method of birth control considered acceptable by the study physician. Contraceptive measures will be reviewed with female subjects at each visit. Dual methods of contraception must be used for 1 month prior to the start of treatment and 6 months after treatment discontinuation.
* A serum pregnancy test obtained at Screen Visit prior to the initiation of treatment must be negative.
* Confirmation by the principal investigator or a sub-investigator that sexually active male subjects are practicing a method of contraception considered acceptable (vasectomy, condom plus spermicide, plus relationship with a female partner who practices an acceptable method of contraception). Contraception must be used during the treatment period and for seven months (or 6 months, according to local label) after the completion of therapy, including condom use by male subjects with pregnant partners.
* For subjects with a history of hypertension or diabetes, written clearance from an ophthalmologist has to be obtained prior to treatment start.

Exclusion Criteria:

* Pregnant women, women who plan to become pregnant, male subjects whose partner wants to become pregnant, and breastfeeding women.
* Previous treatment for chronic hepatitis C with an antiviral or immunomodulating agent or with some interferon or ribavirin product, whether alone or in combination.
* Subjects weighing over 125 kg.
* Suspected hypersensitivity to any interferon or ribavirin product.
* Participation in other clinical trial within 30 days prior to screen into this study.
* Coinfection with hepatitis B virus (HBV), human immunodeficiency virus (HIV), or both.
* Any cause of liver disease other than chronic hepatitis C, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Non-alcoholic steatohepatitis (NASH)
  * Drug-related liver disease
* Active malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma).
* Known coagulation diseases such as hemophilia; hemoglobin diseases (e.g. thalassemia).
* Known glucose 6-phosphate dehydrogenase (G6PD) deficiency
* Evidence of advanced liver disease such as history or presence of ascites, bleeding varices, or hepatic encephalopathy.
* Subjects with organ transplants, except for corneal or hair transplant.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of study, such as:

  * Preexisting psychiatric condition, especially moderate to severe depression, or a history of severe psychiatric disorder, such as psychosis, suicidal ideation, or suicide attempts. Severe depression includes the following:

    * Hospitalization for depression
    * Electroconvulsive therapy for depression, or
    * Depression causing a prolonged absence from work or significantly altering daily functions.
  * Subjects with mild depression may be considered for entry into the study provided that a pre-treatment assessment demonstrates that the subject's emotional status is clinically stable, in which case a management plan must be formulated for the subject; this management plan will become a part of the subject's medical record.
  * Craniocerebral trauma which is not a concussion, or active seizure disorders requiring medication.
  * Clinically significant electrocardiogram (ECG) abnormalities and/or cardiovascular dysfunction within 6 previous months (e.g., angina, congestive heart failure, recent myocardial infarction, or significant arrhythmia).
  * Chronic lung disease (e.g., chronic obstructive lung disease)
  * Poorly controlled diabetes mellitus
  * Immune-mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis)
  * Clinical gout
* Subject is or was a substance abuser, such as alcohol (80 g/day or more), methadone, intravenous(IV), oral or inhaled drugs. To be considered for inclusion into the protocol, the subject must have abstained and agree to abstain from using any of the above for at least 6 months. Subjects treated with buprenorphine (Subutex) who have been stable for 6 months may be included.
* Cirrhotic subjects whose ultrasound confirms hepatocellular carcinoma.
* Any other condition that, in the investigator's opinion, could determine that subject's participation in the study is not indicated or could interfere with the subject's participation in and completion of study.
* Subjacent disease that potentially would require systematic administration of steroids
* Insulin dependent diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Buti M, Lurie Y, Zakharova NG, Blokhina NP, Horban A, Teuber G, Sarrazin C, Balciuniene L, Feinman SV, Faruqi R, Pedicone LD, Esteban R; SUCCESS Study Investigators. Randomized trial of peginterferon alfa-2b and ribavirin for 48 or 72 weeks in patients with hepatitis C virus genotype 1 and slow virologic response. Hepatology. 2010 Oct;52(4):1201-7. doi: 10.1002/hep.23816. PMID 20683847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1428 patients enrolled; 159 patients qualified as slow responders per treatment week 12 and 24 protocol-specified eligibility criteria; 159 patients were randomized
Groups:
- Standard Therapy (48-week Treatment): Slow responders (defined as being polymerase chain reaction [PCR] positive at Week 12 with at least 2 log reduction in viral load and PCR negative at Week 24) who are randomized at Week 48 to stop treatment at Week 48.
- Extended Therapy (72-week Treatment): Slow responders (defined as being PCR positive at Week 12 with at least 2 log reduction in viral load and PCR negative at Week 24) who are randomized at Week 48 to continue treatment to Week 72.
Period: Overall Study
Arm/Group | Standard Therapy (48-week Treatment) | Extended Therapy (72-week Treatment)
Started | 86 | 73
Completed | 78 | 56
Not Completed | 8 | 17
Not completed — Adverse Event | 3 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Protocol Violation | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Administrative | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy (48-week Treatment) | Extended Therapy (72-week Treatment) | Total
Number analyzed (Participants) | 86 | 73 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (9.9) | 46.5 (11.6) | 45.35 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 52 | 46 | 98

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response, Defined as a Plasma HCV-RNA (Hepatitis C Ribonucleic Acid) Level Below the LLQ (Lower Level of Quantitation) at 24 Weeks Post-treatment.
Description: LLQ = 30 IU/mL by reverse transcription polymerase chain reaction (RT-PCR) (Taqman Roche)
Time Frame: 48 or 72 weeks of treatment plus 24 weeks of follow-up.
Population: According to the protocol, the efficacy analysis was carried out on all slow responders (ie, patients who had at least 2 log drop in HCV-RNA level at treatment week 12, and undetectable HCV-RNA at treatment week 24).
Measure: Number; unit: Participants
Arm/Group | Standard Therapy (48-week Treatment) | Extended Therapy (72-week Treatment)
Number analyzed (Participants) | 86 | 73
Participants | 37 | 35
Statistical Analysis 1: Comparison: Standard Therapy (48-week Treatment) vs Extended Therapy (72-week Treatment); Test type: Superiority or Other; p = 0.6445, Asymptotic Z-test; SVR Rate Difference = -4.9, 95% CI [-20.4 to 10.6]

ADVERSE EVENTS:
Arm/Group | Standard Therapy (48-week Treatment)
Serious Adverse Events (participants affected / at risk) | 93/1427
Other Adverse Events (participants affected / at risk) | 1337/1427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (48-week Treatment) (N=1427)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 2 (2)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
THYROIDITIS SUBACUTE (Endocrine disorders) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1)
RETINAL TEAR (Eye disorders) | 1 (1)
VISUAL DISTURBANCE (Eye disorders) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
INTUSSUSCEPTION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (4)
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 4 (5)
PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 1 (1)
ABSCESS ORAL (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 4 (4)
CELLULITIS (Infections and infestations) | 2 (2)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1)
INJECTION SITE ABSCESS (Infections and infestations) | 1 (1)
INJECTION SITE CELLULITIS (Infections and infestations) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1)
ORCHITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 4 (4)
PULMONARY TUBERCULOSIS (Infections and infestations) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SYPHILIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 1 (1)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1)
MULTIPLE DRUG OVERDOSE INTENTIONAL (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ARTERIOGRAM (Investigations) | 1 (1)
HEART RATE INCREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (2)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
UNEQUAL LIMB LENGTH (Musculoskeletal and connective tissue disorders) | 1 (1)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CAROTID ARTERY DISSECTION (Nervous system disorders) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1)
PARKINSONISM (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 3 (3)
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1)
ALCOHOLISM (Psychiatric disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 2 (2)
DELIRIUM (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 4 (4)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1)
HOMICIDAL IDEATION (Psychiatric disorders) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 2 (2)
PARANOIA (Psychiatric disorders) | 2 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 2 (2)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 3 (3)
OLIGURIA (Renal and urinary disorders) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OBLITERATIVE BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1)
ANAL FISSURE EXCISION (Surgical and medical procedures) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (48-week Treatment) (N=1427)
ANAEMIA (Blood and lymphatic system disorders) | 197 (260)
ERYTHROPENIA (Blood and lymphatic system disorders) | 74 (96)
LEUKOPENIA (Blood and lymphatic system disorders) | 183 (268)
NEUTROPENIA (Blood and lymphatic system disorders) | 281 (464)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 94 (112)
DIARRHOEA (Gastrointestinal disorders) | 129 (152)
DRY MOUTH (Gastrointestinal disorders) | 75 (75)
NAUSEA (Gastrointestinal disorders) | 254 (301)
ASTHENIA (General disorders) | 402 (458)
CHILLS (General disorders) | 153 (204)
FATIGUE (General disorders) | 338 (412)
INFLUENZA LIKE ILLNESS (General disorders) | 599 (843)
INJECTION SITE ERYTHEMA (General disorders) | 143 (152)
IRRITABILITY (General disorders) | 157 (169)
PYREXIA (General disorders) | 421 (834)
HAEMOGLOBIN DECREASED (Investigations) | 161 (215)
NEUTROPHIL COUNT DECREASED (Investigations) | 106 (171)
WEIGHT DECREASED (Investigations) | 150 (169)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 77 (112)
ANOREXIA (Metabolism and nutrition disorders) | 156 (160)
DECREASED APPETITE (Metabolism and nutrition disorders) | 103 (107)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 195 (235)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 91 (106)
MYALGIA (Musculoskeletal and connective tissue disorders) | 274 (417)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 77 (81)
DIZZINESS (Nervous system disorders) | 115 (128)
HEADACHE (Nervous system disorders) | 408 (569)
DEPRESSION (Psychiatric disorders) | 139 (156)
INSOMNIA (Psychiatric disorders) | 178 (194)
COUGH (Respiratory, thoracic and mediastinal disorders) | 195 (213)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 111 (124)
ALOPECIA (Skin and subcutaneous tissue disorders) | 318 (328)
DRY SKIN (Skin and subcutaneous tissue disorders) | 188 (199)
PRURITUS (Skin and subcutaneous tissue disorders) | 267 (290)
RASH (Skin and subcutaneous tissue disorders) | 177 (211)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less